CLINICAL TRIAL: NCT02635750
Title: A Study to Investigate the Pharmacokinetic Drug-drug Interaction Following Oral Administration of BI 409306 and Donepezil in Healthy Male and Female Subjects
Brief Title: Investigation of Pharmacokinetic Drug-drug Interaction of BI 409306 and Donepezil in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1289.24; 2015-001694-40 (EudraCT Number)
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306; Donepezil

ARMS (3):
- Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg donepezil (T1) (Experimental): Subjects received treatment in a fixed sequence. First BI 409306 as reference treatment (R1)), then BI 409306 + donepezil as test treatment (T1)).
  Interventions: Drug: BI 409306; Drug: Donepezil
- Part 2: 5 mg donepezil (R2) / 5 mg donepezil + 100 mg BI 409306 (T2) (Experimental): Subjects received first the reference treatment (R2) followed by a washout period, followed by the test treatment (T2).
  Interventions: Drug: BI 409306; Drug: Donepezil
- Part 2: 5 mg donepezil + 100 mg BI 409306 (T2) / 5 mg donepezil (R2) (Experimental): Subjects received first the test treatment 2 (T2) followed by a washout period, followed by the reference treatment 2 (R2)).
  Interventions: Drug: BI 409306; Drug: Donepezil

INTERVENTIONS:
Drug: BI 409306
Drug: Donepezil

SUMMARY:
Part I:

To investigate whether and to what extent donepezil affects single dose pharmacokinetics of BI 409306

Part II:

To investigate whether and to what extent BI 409306 affects the single dose pharmacokinetics of donepezil

ELIGIBILITY:
Inclusion criteria:

* Healthy male/female subjects,
* age of 18 to 55 years,
* body mass index (BMI) of 18.5 to 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:
* Use of adequate contraception, e.g. any of the following methods plus condom:

intrauterine device (non-hormonal)

* Sexually abstinent
* A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy)
* Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 60 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker
* Alcohol abuse Further exclusion criteria apply

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part I (18 subjects entered) of this trial was performed as a one fixed sequence, open-label trial; single doses of BI 409306 and multiple doses of donepezil were administered. Part II (14 subjects entered) was performed as a randomised, open-label, 2-way crossover trial; single doses of donepezil and multiple doses of BI 409306 were administered.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
  Removal of individual subjects if the subject withdrew consent for trial treatment or trial participation, without the need to justify the decision.
Groups:
- Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1): This arm is used in part 1 of this trial only. The subjects received the treatments in a fixed sequence: Reference treatment (R1) / test treatment (T1). The test treatment (T1) was administered after preceding treatment with donepezil for 21 days.
  On day 1 of period 1, one film-coated tablet of 25 milligram (mg) BI 409306 was administered as single oral dose with 240 milliliter (mL) of water after a standardized dinner (R1).
  In period 2, day 1 to 7, subjects received one film-coated tablet of 5 mg donepezil administered orally once daily, followed by 2 film-coated tablets of 5 mg (total: 10 mg) donepezil once daily on day 8 to 21 (up-titration regime).
  On day 1 of period 3, one film-coated tablet of 25 mg BI 409306 was administered as single oral dose together with 2 film-coated tablets of 5 mg (total: 10 mg) donepezil with 240 mL of water after a standardized dinner (T1). There was no washout periods between the visits.
- Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2): This arm is used in part 2 of this trial only. Each subject received first the reference treatment (R2) followed by a washout period of at least 25 days, followed by the test treatment (T2). On day 1 of period 1, one film-coated tablet of 5 mg donepezil (R2) was administered as single oral dose with 240 mL of water in the morning in fasted state, followed by a washout period of at least 25 days. On day 1 of period 2, one film-coated tablet of 5 mg donepezil together with 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 (T2) were administered orally with 240 ml of water in the morning in fasted state. From day 2 to day 7 in period 2, subjects were administered 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 orally once daily.
- Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2): This arm is used in part 2 of this trial only. Each subject received first the test treatment (T2) followed by a washout period of at least 25 days, followed by the reference treatment (R2).
  On day 1 of period 1, one film-coated tablet of 5 mg donepezil together with 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 (T2) were administered orally with 240 ml of water in the morning in fasted state. From day 2 to day 7 in period 1, subjects were administered 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 orally once daily, followed by a washout period of 25 days. On day 1 of period 2, one film-coated tablet of 5 mg donepezil (R2) was administered as single oral dose with 240 mL of water in the morning in fasted state.
Period: Part 1, Period 1
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 18 | 0 | 0
Completed | 18 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 1, Period 2
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 18 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Part 1, Period 3
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 17 | 0 | 0
Completed | 17 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 2, Period 1
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 0 | 7 | 7
Completed | 0 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Part 2, Washout
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 0 | 7 | 7
Completed | 0 | 7 | 7
Not Completed | 0 | 0 | 0
Period: Part 2, Period 2
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2)
Started | 0 | 7 | 7
Completed | 0 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were documented to have received at least 1 dose of trial drug. All 32 subjects of both trial parts were included in the TS. This subject set was used for the safety analysis and presentation of demographic and baseline characteristics and disposition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 25 mg BI 409306 (R1) / 25 mg BI 409306 + 10 mg Donepezil (T1) | Part 2: 5 mg Donepezil (R2) / 5 mg Donepezil + 100 mg BI 409306 (T2) | Part 2: 5 mg Donepezil + 100 mg BI 409306 (T2) / 5mg Donepezil (R2) | Total
Number analyzed (Participants) | 18 | 7 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (8.9) | 45.1 (8.8) | 36.9 (6.3) | 42.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 2 | 15
  Male | 9 | 3 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Part 1: AUC0-tz of BI 409306
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 to the last quantifiable data point.
Time Frame: Within 3 hours (h) prior to administration of BI 409306 and 10, 20, 30, 45 minutes (min) and 1, 1:30, 2:00, 2:30, 3, 4, 5, 6, 8, 10, 12, 14, 16 hours thereafter.
Population: Pharmacokinetic analysis set (PKS) included all subjects who were documented to have taken at least one dose of trial drug and provided at least one pharmacokinetic (PK) parameter that was defined as primary or secondary endpoint and was judged as PK evaluable and not affected by protocol violations. Only participants with non-missing results are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol (nmol)*hour (h)/Litre (L)
Groups:
- 25 mg BI 409306: One film-coated tablet of 25 milligram (mg) BI 409306 was administered as single oral dose with 240 milliliter (mL) of water after a standardized dinner (reference treatment 1 (R1)).
- 25 mg BI 409306 + 10 mg Donepezil: One film-coated tablet of 25 mg BI 409306 was administered as single oral dose together with 2 film-coated tablets of 5 mg (total: 10 mg) donepezil with 240 mL of water after a standardized dinner (test treatment 1 (T1)).
Arm/Group | 25 mg BI 409306 | 25 mg BI 409306 + 10 mg Donepezil
Number analyzed (Participants) | 18 | 17
nanomol (nmol)*hour (h)/Litre (L) | 603 (95.4) | 643 (86.2)
Statistical Analysis 1: Comparison: 25 mg BI 409306 vs 25 mg BI 409306 + 10 mg Donepezil; The statistical model used for the analysis of those endpoints was an analysis of variance (ANOVA) model on the logarithmic scale (natural logarithm). This model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subjects' was considered as random, whereas the other effect was considered as fixed. Abbreviations used: geometric mean (gMean), donepezil (don); Test type: Other; Adjusted gMean ratio(%) = 99.95, 90% CI 2-sided [89.502 to 111.62] — Ratio of BI 409306 25mg with donepezil 10mg and BI 409306 25mg alone (BI 409306+ don / BI 409306). Intra-individual coefficient of variation (gCV (%)) = 18.6

2. Primary Outcome: Part 1: Cmax of BI 409306
Description: Maximum measured concentration of the BI 409306 in plasma.
Time Frame: Within 3 hours (h) prior to administration of BI 409306 and 10, 20, 30, 45 minutes (min) and 1, 1:30, 2:00, 2:30, 3, 4, 5, 6, 8, 10, 12, 14,16 hours thereafter.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 25 mg BI 409306 | 25 mg BI 409306 + 10 mg Donepezil
Number analyzed (Participants) | 18 | 17
nmol/L | 268 (86.2) | 286 (47.8)
Statistical Analysis 1: Comparison: 25 mg BI 409306 vs 25 mg BI 409306 + 10 mg Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted gMean ratio(%) = 100.82, 90% CI 2-sided [81.861 to 124.17] — Ratio of BI 409306 25mg with donepezil 10mg and BI 409306 25mg alone (BI 409306+don / BI 409306). Intra-individual coefficient of variation (gCV (%)) = 35.8

3. Primary Outcome: Part 2: AUC0-tz of Donepezil
Description: Area under the concentration-time curve of donepezil in plasma over the time interval from 0 to the last quantifiable data point.
Time Frame: At approximate 2 hours (h) prior to first administration of donepezil and 1, 2, 2:30, 3, 3:30, 4, 6, 8, 10, 12, 15, 24:30, 48:30, 72:30, 96:30, 120:30, 144:30, 168:30 hours thereafter.
Population: Pharmacokinetic analysis set (PKS) included all subjects who were documented to have taken at least one dose of trial drug and provided at least one pharmacokinetic (PK) parameter that was defined as primary or secondary endpoint and was judged as PK evaluable and not affected by protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*h/ millilitre (mL)
Groups:
- 5 mg Donepezil: One film-coated tablet of 5 mg donepezil (reference treatment 2 (R2)) was administered as single oral dose with 240 mL of water in the morning in fasted state.
- 5 mg Donepezil + 100 mg BI 409306: One film-coated tablet of 5 mg donepezil together with 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 (test treatment 2 (T2)) were administered orally with 240 ml of water in the morning in fasted state on day 1. From day 2 to day 7, subjects were administered 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 orally once daily.
Arm/Group | 5 mg Donepezil | 5 mg Donepezil + 100 mg BI 409306
Number analyzed (Participants) | 14 | 14
nanogram (ng)*h/ millilitre (mL) | 299 (20.4) | 301 (20.6)
Statistical Analysis 1: Comparison: 5 mg Donepezil vs 5 mg Donepezil + 100 mg BI 409306; The PK endpoints were log transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'periods' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Abbreviations used: geometric mean (gMean), donepezil (don); Test type: Other; Adjusted gMean ratio (%) = 100.84, 90% CI 2-sided [97.584 to 104.19] — Ratio of donepezil 5mg with BI 409306 100mg and donepezil 5mg alone (BI 409306+don / don). Intra-individual coefficient of variation (gCV (%)) = 4.9

4. Primary Outcome: Part 2: Cmax of Donepezil
Description: Maximum measured concentration of the donepezil in plasma.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 5 mg Donepezil | 5 mg Donepezil + 100 mg BI 409306
Number analyzed (Participants) | 14 | 14
ng/mL | 6.23 (27.5) | 7.04 (30.0)
Statistical Analysis 1: Comparison: 5 mg Donepezil vs 5 mg Donepezil + 100 mg BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted gMean ratio(%) = 113.08, 90% CI 2-sided [106.41 to 120.15] — Ratio of donepezil 5mg with BI 409306 100mg and donepezil 5mg alone. (BI 409306+don / don) Intra-individual coefficient of variation (gCV (%)) = 9.0

5. Secondary Outcome: Part 1: AUC 0-infinity of BI 409306
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: At approximate 3 hours (h) prior to administration of BI 409306 and 10, 20, 30, 45 minutes (min) and 1, 1:30, 2:00, 2:30, 3, 4, 5, 6, 8, 10, 12, 14,16 hours thereafter.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 25 mg BI 409306 | 25 mg BI 409306 + 10 mg Donepezil
Number analyzed (Participants) | 18 | 17
nmol*h/L | 604 (95.5) | 644 (86.4)
Statistical Analysis 1: Comparison: 25 mg BI 409306 vs 25 mg BI 409306 + 10 mg Donepezil; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted gMean ratio(%) = 100.01, 90% CI 2-sided [89.549 to 111.68] — Ratio of BI 409306 25mg with donepezil 10mg and BI 409306 25mg alone (BI 409306+don/ BI 409306). Intra-individual coefficient of variation (gCV(%)) = 18.6

6. Secondary Outcome: Part 2: AUC0-infinity of Donepezil
Description: This outcome measure presents the area under the concentration-time curve of donepezil in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 5 mg Donepezil +100 mg BI 409306: One film-coated tablet of 5 mg donepezil together with 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 (test treatment 2 (T2)) were administered orally with 240 ml of water in the morning in fasted state on day 1. From day 2 to day 7, subjects were administered 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 orally once daily.
Arm/Group | 5 mg Donepezil | 5 mg Donepezil +100 mg BI 409306
Number analyzed (Participants) | 14 | 14
ng*h/mL | 386 (29.9) | 380 (23.4)
Statistical Analysis 1: Comparison: 5 mg Donepezil vs 5 mg Donepezil +100 mg BI 409306; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted gMean ratio(%) = 98.38, 90% CI 2-sided [93.413 to 103.60] — Ratio of donepezil 5mg with BI 409306 100mg and donepezil 5mg alone (BI 409306+don / don). Intra-individual coefficient of variation (gCV (%)) = 7.7

ADVERSE EVENTS:
Time Frame: From first drug intake until end of the residual effect period (REP), which was defined as 24 hours after last intake of BI 409306 or 14 days after last donepezil (DON) administration. In case of combined treatment period started from first combined drug intake until last combined drug intake plus 14 days (REP of DON). Up to 1 day for 'Part 1: 25 mg BI'; up to 14 days for 'Part 1: 25mg BI+ 10mg DON', 'Part 2: 5mg DON' and 'Part 2: 5mg DON+ 100mg BI' and up to 21 days for 'Part 1: 5mg/10mg DON'.
Description: The treated set (TS) included all subjects who were documented to have received at least 1 dose of trial drug.
Groups:
- Part 1: 25 mg BI 409306: One film-coated tablet of 25 milligram (mg) BI 409306 was administered as single oral dose with 240 milliliter (mL) of water after a standardized dinner (reference treatment 1 (R1)).
- Part 1: 5 mg Donepezil /10 mg Donepezil: Period 2: On day 1 to 7, subjects received one film-coated tablet of 5 mg donepezil administered orally once daily, followed by 2 film-coated tablets of 5 mg (total: 10 mg) donepezil once daily on day 8 to 21.
- Part 1: 25 mg BI 409306 25mg + 10 mg Donepezil: Period 3: One film-coated tablet of 25 mg BI 409306 was administered as single oral dose together with 2 film-coated tablets of 5 mg (total: 10 mg) donepezil with 240 mL of water after a standardized dinner (test treatment 1 (T1)).
- Part 2: 5 mg Donepezil: One film-coated tablet of 5 mg donepezil (reference treatment 2 (R2)) was administered as single oral dose with 240 mL of water in the morning in fasted state.
- Part 2: 5mg Donepezil + 100 mg BI 409306: One film-coated tablet of 5 mg donepezil together with 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 (test treatment 2 (T2)) were administered orally with 240 ml of water in the morning in fasted state on day 1. From day 2 to day 7, subjects were administered 4 film-coated tablets of 25 mg (total: 100 mg) BI 409306 orally once daily.
Arm/Group | Part 1: 25 mg BI 409306 | Part 1: 5 mg Donepezil /10 mg Donepezil | Part 1: 25 mg BI 409306 25mg + 10 mg Donepezil | Part 2: 5 mg Donepezil | Part 2: 5mg Donepezil + 100 mg BI 409306
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/18 | 15/18 | 5/17 | 4/14 | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 25 mg BI 409306 (N=18) | Part 1: 5 mg Donepezil /10 mg Donepezil (N=18) | Part 1: 25 mg BI 409306 25mg + 10 mg Donepezil (N=17) | Part 2: 5 mg Donepezil (N=14) | Part 2: 5mg Donepezil + 100 mg BI 409306 (N=14)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 4
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 5
Vision blurred (Eye disorders) | 0 | 3 | 0 | 0 | 0
Visual brightness (Eye disorders) | 2 | 0 | 0 | 0 | 3
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 10 | 2 | 1 | 4
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 1 | 1
Vessel puncture site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 10 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 3 | 1 | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.